CLINICAL TRIAL: NCT00006968
Title: Non-Myeloablative Chemotherapy Followed By Related Allogeneic Stem Cell Rescue In Patients With Advanced Renal Cell Carcinoma
Brief Title: Pentostatin Followed by Peripheral Stem Cell Transplantation in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068349; UCLA-0001032; SUPERGEN-UCLA-000103201; NCI-G00-1879
Record Dates: First submitted 2000-12-06; First posted 2003-06-27 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Filgrastim; Cyclosporine; Pentostatin; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: cyclosporine
Drug: pentostatin
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with donor peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of pentostatin followed by peripheral stem cell transplantation in treating patients who have advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the duration and efficiency of hematopoietic and immunologic engraftment in patients with advanced renal cell carcinoma treated with pentostatin followed by related allogeneic stem cell transplantation.
* Determine the hematologic and non-hematologic toxic effects of this regimen in these patients.
* Determine the incidence and severity of graft-versus-host disease in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of pentostatin.

* Phase I: Patients receive pentostatin IV on days -7, -5, and -3 followed by allogeneic stem cell transplantation on day 0. Beginning on day 1, patients receive filgrastim (G-CSF) IV over 1 hour or subcutaneously daily until blood counts recover. As graft-versus-host disease prophylaxis, patients receive cyclosporine IV continuously until stem cell engraftment and then orally with gradual tapering.

Cohorts of 3 to 6 patients receive escalating doses of pentostatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive treatment as in phase I at the MTD for pentostatin. Patients are followed weekly for 60 days and then monthly for 10 months.

PROJECTED ACCRUAL: A total of 24 patients (12 per phase) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced renal cell cancer
* No bone metastases
* No CNS disease
* Must have an allogeneic donor available

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-1

Life expectancy:

* 3 to 6 months

Hematopoietic:

* Hemoglobin at least 10 g/dL
* Complete blood count normal

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* Transaminases no greater than 4 times ULN
* No evidence of portal hypertension

Renal:

* Creatinine no greater than 2.0 mg/dL
* No uncontrolled hypercalcemia

Cardiovascular:

* No New York Heart Association class 3 or 4 heart disease

Pulmonary:

* DLCO at least 40% of predicted

Other:

* No severe functional neurological impairment
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior biologic therapy

Chemotherapy:

* No more than 6 months of prior chemotherapy

Endocrine therapy:

* At least 1 year since prior steroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2000-09; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary J. Schiller, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States